CLINICAL TRIAL: NCT05577702
Title: A Randomized, Open-Label, Multicenter, Phase 2, Umbrella Study to Evaluate the Preliminary Efficacy, Safety, and Pharmacodynamics of Tislelizumab Monotherapy and Multiple Tislelizumab-based Immunotherapy Combinations With and Without Chemotherapy as Neoadjuvant Treatment in Chinese Patients With Resectable Stage II to IIIA Non-Small Cell Lung Cancer
Brief Title: Efficacy, Safety, and Pharmacodynamics of Tislelizumab Monotherapy and Multiple Tislelizumab-based Immunotherapy Combinations in Participants With Resectable Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-LC-202; CTR20222760 (Other: ChinaDrugTrials)
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Cisplatin; Carboplatin; Pemetrexed; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm 1A: Tislelizumab Monotherapy (Experimental): Participants with tumor programmed death protein ligand-1 (PD-L1) expression ≥ 50% received 200 mg tislelizumab intravenously once every 3 weeks for 2-4 cycles followed by surgical removal of the tumor.
  Interventions: Drug: Tislelizumab
- Arm 1B: Tislelizumab + Ociperlimab (Experimental): Participants with tumor PD-L1 expression ≥ 50% received 200 mg tislelizumab and 900 mg ociperlimab intravenously once every 3 weeks for 2-4 cycles followed by surgical removal of the tumor.
  Interventions: Drug: Tislelizumab; Drug: Ociperlimab
- Arm 1C: Alcestobart + Tislelizumab (Experimental): Participants with tumor PD-L1 expression ≥ 50% received 200 mg tislelizumab and 600 mg alcestobart intravenously once every 3 weeks for 2-4 cycles followed by surgical removal of the tumor.
  Interventions: Drug: Tislelizumab; Drug: Alcestobart
- Arm 2A: Tislelizumab and Chemotherapy (Experimental): Participants with tumor PD-L1 expression < 50% received 200 mg tislelizumab and chemotherapy consisting of cisplatin or carboplatin with either pemetrexed or paclitaxel administered intravenously once every 3 weeks for 2-4 cycles followed by surgical removal of the tumor.
  Interventions: Drug: Tislelizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel
- Arm 2C: Alcestobart + Tislelizumab + Chemotherapy (Experimental): Participants with tumor PD-L1 expression < 50% received 200 mg tislelizumab, 600 mg alcestobart and chemotherapy consisting of cisplatin or carboplatin with either pemetrexed or paclitaxel administered intravenously once every 3 weeks for 2-4 cycles followed by surgical removal of the tumor.
  Interventions: Drug: Tislelizumab; Drug: Alcestobart; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Drug: Paclitaxel

INTERVENTIONS:
Drug: Tislelizumab — Administered as an intravenous infusion once every 3 weeks
  Other Names: BGB-A317; Tevimbra
Drug: Ociperlimab — Administered as an intravenous infusion once every 3 weeks
  Other Names: BGB-A1217
  Arms: Arm 1B: Tislelizumab + Ociperlimab
Drug: Alcestobart — Administered as an intravenous infusion once every 3 weeks
  Other Names: LBL-007
  Arms: Arm 1C: Alcestobart + Tislelizumab; Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Drug: Cisplatin — 75 mg/m^2 administered as an intravenous infusion once every 3 weeks
  Arms: Arm 2A: Tislelizumab and Chemotherapy; Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Drug: Carboplatin — Administered as an intravenous infusion once every 3 weeks at an area under the curve (AUC) of 5 mg/mL/min
  Arms: Arm 2A: Tislelizumab and Chemotherapy; Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Drug: Pemetrexed — 500 mg/m^2 administered as an intravenous infusion once every 3 weeks in participants with non-squamous NSCLC
  Arms: Arm 2A: Tislelizumab and Chemotherapy; Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Drug: Paclitaxel — 175 mg/m^2 administered as an intravenous infusion once every 3 weeks in participants with squamous NSCLC
  Arms: Arm 2A: Tislelizumab and Chemotherapy; Arm 2C: Alcestobart + Tislelizumab + Chemotherapy

SUMMARY:
This study was conducted to evaluate the preliminary effectiveness and safety of treatment with tislelizumab alone and in combination with other investigational agents prior to surgery (neoadjuvant treatment) in adults with non-small cell lung cancer (NSCLC) that is able to be removed by surgery.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter, Phase 2, umbrella study to evaluate the preliminary efficacy, safety, and pharmacodynamics of tislelizumab as monotherapy and in combination with investigational agents as neoadjuvant treatment in Chinese participants with resectable Stage II to IIIA NSCLC. The study is designed with the flexibility of adding treatment arms as new treatments become available or discontinuing treatment arms that demonstrate minimal clinical activity or unacceptable toxicity, and of modifying the participant population.

The study consisted of a neoadjuvant treatment phase (2 - 4 cycles of treatment), a surgery phase and a follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1
* Histologically confirmed Stage II-IIIA NSCLC (per the Eighth American Joint Committee on Cancer/Union Internationale Contre le Cancer [NSCLC] staging system)
* Evaluation by an attending thoracic surgeon to confirm eligibility for an R0 resection with curative intent
* Adequate hematologic and organ function, defined by protocol-specified laboratory test results, obtained ≤ 7 days before randomization
* Provide formalin-fixed paraffin-embedded block (preferred) or at least 15 freshly cut unstained FFPE slides of the primary tumor for biomarker evaluation during screening

Exclusion Criteria:

* Any prior antineoplastic therapy(ies) for current lung cancer (eg, radiotherapy, targeted therapies, ablation, or other systemic or local antineoplastic treatment)
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, anti-cell immunoglobulin and ITIM domain (TIGIT), anti-lymphocyte activation gene-3 (LAG-3), or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Has mixed small cell lung cancer
* Participants with large cell neuroendocrine carcinoma (LCNEC)
* The presence of locally advanced unresectable NSCLC regardless of stage or metastatic disease
* Known epidermal growth factor receptor (EGFR) sensitizing mutations and/or anaplastic lymphoma kinase (ALK) rearrangement

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (14):
- China (14):
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Guangzhou Medical Universitydatansha Hospital), Guangzhou, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Anyang Cancer Hospital, Anyang, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University Branch Xianghu, Nanchang, Jiangxi
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Hwa Mei Hospital, University of Chinese Academy of Sciences (Ningbo No Hospital), Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Begene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  Beigene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for Beigene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 121 participants at study sites in China.
Pre-assignment Details: In Substudy 1 participants with programmed death-ligand 1 (PD-L1) expression ≥ 50% were randomized to 1 of 3 treatment groups in a 1:1:1 ratio.
  In Substudy 2 participants with PD-L1 expression < 50% were randomized into 1 of 2 treatment groups in a 1:2 ratio.
Groups:
- Arm 2C: Alcestobart + Tislelizumab + Chemotherapy: Participants with tumor PD-L1 expression < 50% received 200 mg tislelizumab, 600 mg alcestobart and chemotherapy consisting of cisplatin or carboplatin with either pemetrexed or paclitaxel administered intravenously once every 3 weeks for 2 - 4 cycles followed by surgical removal of the tumor.
Period: Overall Study
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Started | 20 | 20 | 20 | 20 | 41
Treated | 20 | 20 | 20 | 19 | 40
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 20 | 20 | 20 | 20 | 41
Not completed — Study Ended by Sponsor | 19 | 17 | 19 | 16 | 38
Not completed — Death | 1 | 2 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1A: Tislelizumab Monotherapy: Participants with tumor PD-L1 expression ≥ 50% received 200 mg tislelizumab intravenously once every 3 weeks for 2 - 4 cycles followed by surgical removal of the tumor.
- Total: Total of all reporting groups
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 41 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (6.68) | 63.1 (6.78) | 62.7 (8.03) | 61.0 (6.86) | 61.9 (9.76) | 62.3 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 3 | 10 | 19
  Male | 18 | 19 | 17 | 17 | 31 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 20 | 20 | 41 | 121
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 20 | 20 | 20 | 20 | 41 | 121
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG Performance Scale is used to assess a patient's disease status. 0 = Fully active, able to carry out all pre-disease performance without restriction;
  1. = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  2. = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours;
  3. = Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  4. = Completely disabled, confined to bed or chair;
  5. = Dead.
  Participants
    0 (Fully Active) | 9 | 7 | 8 | 9 | 22 | 55
    1 (Ambulatory with Restricted Activities) | 11 | 13 | 12 | 11 | 19 | 66
Smoking Status [Count of Participants; unit: Participants]
  Current | 3 | 1 | 4 | 2 | 5 | 15
  Former | 15 | 15 | 12 | 15 | 22 | 79
  Never | 2 | 4 | 4 | 3 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Major Pathological Response (MPR) Rate
Description: Tumor tissue and lymph node tissue obtained from surgical resection were sent to a central laboratory according to study pathology manuals for pathological response analysis. MPR rate is defined as the percentage of participants with ≤ 10% residual viable tumor in the resected primary tumor and all resected lymph nodes as assessed by blinded independent pathology review (BIPR). Participants without surgery or pathological results were considered non-responders.
Time Frame: At the time of surgery, approximately Week 16
Population: The Intent-to-Treat (ITT) analysis set includes all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 41
percentage of participants | 45.0 [23.1 to 68.5] | 50.0 [27.2 to 72.8] | 40.0 [19.1 to 63.9] | 55.0 [31.5 to 76.9] | 34.1 [20.1 to 50.6]
Statistical Analysis 1: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1B: Tislelizumab + Ociperlimab; Test type: Other; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.35 to 4.24] — Mantel-Haenszel common odds ratio was estimated along with its 95% confidence interval (CI) constructed by a normal approximation of log odds ratio and the Robins, Breslow, and Greenland variance estimate without stratification
Statistical Analysis 2: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1C: Alcestobart + Tislelizumab; Test type: Other; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.23 to 2.86] — Mantel-Haenszel common odds ratio was estimated along with its 95% CI constructed by a normal approximation of log odds ratio and the Robins, Breslow, and Greenland variance estimate without stratification
Statistical Analysis 3: Comparison: Arm 2A: Tislelizumab and Chemotherapy vs Arm 2C: Alcestobart + Tislelizumab + Chemotherapy; Test type: Other; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.14 to 1.26] — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Pathological Complete Response (pCR)
Description: Pathological complete response is defined as the percentage of participants with absence of residual tumor in the resected primary tumor and all resected lymph nodes as assessed by the BIPR. Participants without surgery or pathological results were considered as non-responders.
Time Frame: At the time of surgery, approximately Week 16
Population: Intent to treat analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 41
percentage of participants | 30.0 [11.9 to 54.3] | 30.0 [11.9 to 54.3] | 40.0 [19.1 to 63.9] | 35.0 [15.4 to 59.2] | 17.1 [7.2 to 32.1]
Statistical Analysis 1: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1B: Tislelizumab + Ociperlimab; Test type: Other; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.26 to 3.87] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1C: Alcestobart + Tislelizumab; Test type: Other; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.42 to 5.76] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Arm 2A: Tislelizumab and Chemotherapy vs Arm 2C: Alcestobart + Tislelizumab + Chemotherapy; Test type: Other; Odds Ratio (OR) = 0.38, 95% CI 2-sided [0.11 to 1.30] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the time from randomization until any of the following events, whichever occurred first: radiographic disease progression that precludes definitive surgery, local or distant recurrence as assessed by investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause. Local recurrence is defined as recurrence in the ipsilateral thorax (lymph node or lung on the same side as Baseline location) including lung parenchyma, bronchial stump, main trachea, hilum or mediastinal lymph nodes (including subcarinal lymph nodes), pleura and chest wall diagnosed by radiological examination and/or histopathological confirmation. Distant recurrence (metastasis) is defined as spread of disease beyond the area of the ipsilateral thorax (including contralateral area and other organs) diagnosed by radiological examination and/or histopathological confirmation. Median EFS was estimated using Kaplan-Meier methodology.
Time Frame: From randomization until the end of study, maximum time on study was 22 months in Substudy 1 and 13 months in Substudy 2.
Population: Intent to treat analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 41
months | NA [10.3 to NA] — Could not be estimated due to insufficient number of events | NA [3.7 to NA] — Could not be estimated due to insufficient number of events | 11.4 [11.4 to NA] — Could not be estimated due to insufficient number of events | 11.6 [7.9 to NA] — Could not be estimated due to insufficient number of events | NA [10.9 to NA] — Could not be estimated due to insufficient number of events
Statistical Analysis 1: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1B: Tislelizumab + Ociperlimab; Test type: Other; Hazard Ratio (HR) = 2.54, 95% CI 2-sided [0.46 to 13.94] — Hazard ratio and 95% CIs were estimated using a Cox regression model
Statistical Analysis 2: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1C: Alcestobart + Tislelizumab; Test type: Other; Hazard Ratio (HR) = 2.26, 95% CI 2-sided [0.37 to 13.75] — Hazard ratio and 95% CIs were estimated using a Cox regression model
Statistical Analysis 3: Comparison: Arm 2A: Tislelizumab and Chemotherapy vs Arm 2C: Alcestobart + Tislelizumab + Chemotherapy; Test type: Other; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.28 to 3.52] — Hazard ratio and 95% CIs were estimated using a Cox regression model

4. Secondary Outcome: Event-free Survival Rate
Description: Event-free survival rate is defined as the percentage of participants with none of the following events: radiographic disease progression that precludes definitive surgery, local or distant recurrence as assessed by investigator per RECIST v1.1, or death due to any cause. Local recurrence is defined as recurrence in the ipsilateral thorax (lymph node or lung on the same side as Baseline location) including lung parenchyma, bronchial stump, main trachea, hilum or mediastinal lymph nodes (including subcarinal lymph nodes), pleura and chest wall diagnosed by radiological examination and/or histopathological confirmation. Distant recurrence (metastasis) is defined as spread of disease beyond the area of the ipsilateral thorax (including contralateral area and other organs) diagnosed by radiological examination and/or histopathological confirmation. EFS rates were estimated using the Kaplan-Meier method with the corresponding 95% confidence interval constructed using Greenwood's formula.
Time Frame: 12 months and 24 months after randomization
Population: Intent to treat analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 41
percentage of participants
  12 months | 75.3 [24.5 to 94.4] | 60.0 [17.8 to 86.0] | 44.0 [1.1 to 86.1] | 0.0 [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | 50.5 [15.0 to 78.2]
  24 months | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | 0.0 [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death due to any cause. Median OS was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 3
Population: Intent to treat analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 41
months | NA [NA to NA] — Could not be estimated due to an insufficient number of events | NA [NA to NA] — Could not be estimated due to an insufficient number of events | NA [11.4 to NA] — Could not be estimated due to an insufficient number of events | NA [11.6 to NA] — Could not be estimated due to an insufficient number of events | NA [NA to NA] — Could not be estimated due to an insufficient number of events
Statistical Analysis 1: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1B: Tislelizumab + Ociperlimab; Test type: Other; Hazard Ratio (HR) = 2.29, 95% CI 2-sided [0.21 to 25.30] — Hazard ratio and 95% CIs were estimated using a Cox regression model
Statistical Analysis 2: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1C: Alcestobart + Tislelizumab; Test type: Other; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.06 to 15.89] — Hazard ratio and 95% CIs were estimated using a Cox regression model
Statistical Analysis 3: Comparison: Arm 2A: Tislelizumab and Chemotherapy vs Arm 2C: Alcestobart + Tislelizumab + Chemotherapy; Test type: Other; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.05 to 1.71] — Hazard ratio and 95% CIs were estimated using a Cox regression model

6. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate is defined as the percentage of participants who were still alive at the analysis time points. OS rates were estimated using the Kaplan-Meier method with the corresponding 95% confidence interval constructed using Greenwood's formula.
Time Frame: 12 months and 24 months after randomization
Population: Intent to treat analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 41
percentage of participants
  12 months | 91.7 [53.9 to 98.8] | 89.7 [64.8 to 97.3] | 90.0 [47.3 to 98.5] | 58.6 [8.4 to 89.2] | 94.9 [81.2 to 98.7]
  24 months | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time

7. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS is defined as the time from the first date of no disease (ie, participants who underwent margin-negative [R0] resection) to local or distant recurrence, as assessed by the investigator according to RECIST v1.1, or death due to any cause, whichever occurred first. Median DFS was estimated using Kaplan-Meier methodology.
Time Frame: as for outcome 3
Population: Participants in the intent to treat analysis set with planned surgery who have undergone R0 resection.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 16 | 14 | 12 | 17 | 31
months | NA [8.4 to NA] — Could not be estimated due to an insufficient number of events | NA [8.0 to NA] — Could not be estimated due to an insufficient number of events | NA [8.8 to NA] — Could not be estimated due to an insufficient number of events | 8.7 [4.0 to NA] — Could not be estimated due to an insufficient number of events | NA [9.0 to NA] — Could not be estimated due to an insufficient number of events
Statistical Analysis 1: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1B: Tislelizumab + Ociperlimab; Test type: Other; Hazard Ratio (HR) = 2.88, 95% CI 2-sided [0.26 to 32.37] — Hazard ratio and 95% CIs were estimated using a Cox regression model
Statistical Analysis 2: Comparison: Arm 1A: Tislelizumab Monotherapy vs Arm 1C: Alcestobart + Tislelizumab; Test type: Other; Hazard Ratio (HR) = 1.73, 95% CI 2-sided [0.11 to 27.89] — Hazard ratio and 95% CIs were estimated using a Cox regression model
Statistical Analysis 3: Comparison: Arm 2A: Tislelizumab and Chemotherapy vs Arm 2C: Alcestobart + Tislelizumab + Chemotherapy; Test type: Other; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.19 to 3.27] — Hazard ratio and 95% CIs were estimated using a Cox regression model

8. Secondary Outcome: Disease-free Survival Rate
Description: Disease-free survival rate is defined as the percentage of participants with none of the following events: Local or distant recurrence as assessed by the investigator per RECIST v1.1, or death due to any cause. Local recurrence is defined as recurrence in the ipsilateral thorax (lymph node or lung on the same side as Baseline location) including lung parenchyma, bronchial stump, main trachea, hilum or mediastinal lymph nodes (including subcarinal lymph nodes), pleura and chest wall diagnosed by radiological examination and/or histopathological confirmation. Distant recurrence (metastasis) is defined as spread of disease beyond the area of the ipsilateral thorax (including contralateral area and other organs) diagnosed by radiological examination and/or histopathological confirmation. DFS rates were estimated using the Kaplan-Meier method with the corresponding 95% confidence interval constructed using Greenwood's formula.
Time Frame: 12 months and 24 months after randomization
Population: Participants in the intent to treat analysis set with planned surgery who have undergone R0 resection.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 16 | 14 | 12 | 17 | 31
percentage of participants
  12 months | 75.0 [12.8 to 96.1] | 60.6 [7.5 to 90.8] | 50.0 [0.6 to 91.0] | 0.0 [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time
  24 months | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | 0.0 [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time | NA [NA to NA] — Could not be estimated due to an insufficient number of events and follow-up time

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence that, at any dose:
  * Resulted in death
  * Was life-threatening
  * Required hospitalization or prolongation of existing hospitalization
  * Resulted in disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was considered a significant medical AE by the investigator or sponsor based on medical judgement (eg, may have jeopardized the participant or may require medical/surgical intervention to prevent one of the outcomes listed above).
  Immune-mediated adverse events (imAEs) are autoimmune-mediated complications that may develop in response to immunotherapeutic agents. Immune-mediated AEs were collected from the date of first dose of study drug to 90 days after the last dose of study drug, regardless of whether the participant started a new anticancer therapy or prespecified adjuvant treatment. imAEs were identified by the investigator based on a standard process defined in the Protocol.
Time Frame: From first dose of study drug until 30 days after last dose or new anticancer treatment, whichever occurred first, or up to 90 days after the last dose for imAEs; maximum duration of treatment was 14 weeks.
Population: The safety analysis set included all enrolled participants who received ≥ 1 dose of neoadjuvant treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 20 | 20 | 20 | 19 | 40
Participants
  Any TEAE | 7 | 14 | 15 | 19 | 39
  Serious adverse events | 0 | 3 | 2 | 2 | 13
  Immune-mediated AEs | 0 | 6 | 3 | 2 | 17

10. Secondary Outcome: Feasibility of Surgery
Description: Feasibility of surgery was assessed by the number of participants who underwent surgical resection (surgery) within 6 weeks of last dose of study drug, had delayed or canceled surgery, the approach of surgery, duration of surgery (see next outcome measure) ,and the number of participants who underwent an exploratory thoracotomy, a surgical procedure in which a cut is made between the ribs to see and reach the lungs or other organs in the chest or thorax. Exploratory thoracotomy was not counted as surgery.
Time Frame: At the time of surgery, approximately Week 16
Population: Intent to treat analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 41
Participants
  Underwent Surgery | 16 | 14 | 12 | 17 | 31
  Received open surgery | 4 | 5 | 6 | 4 | 9
  Received minimally invasive surgery | 12 | 9 | 6 | 13 | 22
  Received Exploratory Thoracotomy | 1 | 0 | 0 | 1 | 0
  Delayed Surgery | 7 | 3 | 3 | 2 | 8
  No Surgery or Exploratory Thoracotomy | 3 | 6 | 8 | 1 | 9

11. Secondary Outcome: Duration of Surgery
Description: The duration of surgery is defined as the time interval from the start of the surgical procedure to its completion.
Time Frame: Approximately Week 16
Population: Participants in the intent to treat analysis set who underwent surgery and who had complete records of both surgery start and stop times recorded.
Measure: Median (Full Range); unit: hours
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
Number analyzed (Participants) | 15 | 14 | 12 | 17 | 31
hours | 3.33 [2.5 to 5.3] | 3.50 [2.3 to 5.3] | 3.39 [2.3 to 8.7] | 4.30 [2.7 to 8.0] | 4.05 [2.0 to 6.6]

ADVERSE EVENTS:
Time Frame: Deaths were collected from randomization up to the end of study; maximum time on study was 22 months in Substudy 1 and 13 months in Substudy 2. Adverse events were collected from first dose of study drug until 30 days after last dose or new anticancer treatment, whichever occurred first, or up to 90 days after the last dose for imAEs; maximum duration of treatment was 14 weeks.
Arm/Group | Arm 1A: Tislelizumab Monotherapy | Arm 1B: Tislelizumab + Ociperlimab | Arm 1C: Alcestobart + Tislelizumab | Arm 2A: Tislelizumab and Chemotherapy | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/20 | 2/20 | 1/20 | 3/20 | 2/41
Serious Adverse Events (participants affected / at risk) | 0/20 | 3/20 | 2/20 | 2/19 | 13/40
Other Adverse Events (participants affected / at risk) | 7/20 | 14/20 | 14/20 | 19/19 | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1A: Tislelizumab Monotherapy (N=20) | Arm 1B: Tislelizumab + Ociperlimab (N=20) | Arm 1C: Alcestobart + Tislelizumab (N=20) | Arm 2A: Tislelizumab and Chemotherapy (N=19) | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy (N=40)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myocardial injury (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Pyrexia (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1A: Tislelizumab Monotherapy (N=20) | Arm 1B: Tislelizumab + Ociperlimab (N=20) | Arm 1C: Alcestobart + Tislelizumab (N=20) | Arm 2A: Tislelizumab and Chemotherapy (N=19) | Arm 2C: Alcestobart + Tislelizumab + Chemotherapy (N=40)
Anaemia (Blood and lymphatic system disorders) | 1 (4) | 3 (4) | 4 (7) | 10 (20) | 23 (57)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (11) | 14 (28)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 3 (5)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid disorder (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 7 (9)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 7 (8) | 7 (10)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 3 (3)
Asthenia (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Chest pain (General disorders and administration site conditions) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 5 (8)
Influenza like illness (General disorders and administration site conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (4)
Malaise (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7)
Pain (General disorders and administration site conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders and administration site conditions) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fascioliasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (5) | 4 (4) | 5 (5) | 10 (13)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (6) | 4 (7) | 7 (8) | 10 (19)
Bile acids increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Blood bilirubin increased (Investigations) | 3 (4) | 0 (0) | 1 (2) | 2 (2) | 4 (5)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (6) | 2 (2) | 0 (0) | 2 (5)
Blood homocysteine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Blood iron decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (7)
Blood urea increased (Investigations) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 3 (3)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Glucose urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung diffusion test decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 5 (16)
Myoglobin blood increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 16 (39) | 27 (68)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 5 (6)
Neutrophil percentage decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (5)
Neutrophil percentage increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 6 (6) | 7 (12)
Prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (4)
Serum amyloid A protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 12 (30) | 20 (47)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2)
pH urine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 11 (14)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 3 (7) | 6 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 5 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 3 (3)
Coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 3 (5)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 10 (10)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (2) | 1 (2) | 9 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT05577702/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT05577702/SAP_001.pdf